CLINICAL TRIAL: NCT03446001
Title: Randomized, Double-Blind, Placebo-Controlled, Three-Arm, 12-Month, Safety and Efficacy Study of TRx0237 Monotherapy in Subjects With Alzheimer's Disease Followed by a 12-Month Open-Label Treatment
Brief Title: Safety and Efficacy of TRx0237 in Subjects With Alzheimer's Disease Followed by Open-Label Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-237-039
Expanded Access: NCT03539380 (Available)
Record Dates: First submitted 2018-02-08; First posted 2018-02-26 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — hydromethylthionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TRx0237 16 mg/day (Experimental)
  Interventions: Drug: TRx0237 16 mg/day
- Control (Placebo Comparator)
  Interventions: Drug: Control
- TRx0237 8 mg/day (Experimental)
  Interventions: Drug: TRx0237 8 mg/day

INTERVENTIONS:
Drug: TRx0237 16 mg/day — Oral TRx0237 4-mg tablets administered twice daily
  Arms: TRx0237 16 mg/day
Drug: Control — Oral placebo tablets (some of which contain a urinary discolorant) administered twice daily
  Arms: Control
Drug: TRx0237 8 mg/day — Oral TRx0237 4-mg tablet administered twice daily
  Arms: TRx0237 8 mg/day

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TRx0237 16 mg/day and 8 mg/day in the treatment of subjects with Alzheimer's Disease compared to placebo. In addition, an open-label, delayed-start phase is included to demonstrate a disease-modifying effect of TRx0237.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease (AD), encompassing probable AD and mild cognitive impairment due to AD (MCI-AD) based on the 2011 National Institute on Aging and Alzheimer's Association (NIA/AA) criteria
* Documented PET scan that is positive for amyloid
* Mini-Mental State Examination (MMSE) score of 16-27 (inclusive), subject to stratification requirements
* Global Clinical Dementia Rating (CDR) of 0.5 to 2 (if 0.5, including a score of >0 in one of the functional domains: Community Affairs, Home and Hobbies, or Personal Care)
* Age <90 years
* Females must be surgically sterile, have undergone bilateral tubal occlusion / ligation, be post-menopausal, or use adequate contraception
* Subject, and/or, in the case of reduced decision-making capacity, legally acceptable representative(s) consistent with local and national law is/are able to read, understand, and provide written informed consent in the designated language of the study site
* Has one or more identified adult study partner who either lives with the subject or has sufficient contact to provide assessment of changes in subject behavior and function over time and information on safety and tolerability; is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language(s) at the study site; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study drug
* Must not be taking an acetylcholinesterase inhibitor and/or memantine for at least 60 days at the time of the Baseline assessments
* Able to comply with the study procedures in the view of the Investigator

Exclusion Criteria:

* Significant central nervous system disorder other than probable AD or MCI-AD
* Significant intracranial focal or vascular pathology seen on brain MRI scan that would lead to a diagnosis other than probable AD or MCI-AD
* Clinical evidence or history of cerebrovascular accident; transient ischemic attack; significant head injury, for example, associated loss of consciousness, skull fracture or persisting cognitive impairment; other unexplained or recurrent loss of consciousness for ≥15 minutes
* Epilepsy (a single prior seizure >6 months prior to Screening is considered acceptable)
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria met for major depressive disorder; schizophrenia; other psychotic disorders, bipolar disorder; substance (including alcohol) related disorders
* Metal implants in the head, pacemaker, cochlear implants, or any other non-removable items that are contraindications to MRI
* Resides in hospital or moderate to high dependency continuous care facility
* Any physical disability that would prevent completion of study procedures or assessments
* History of swallowing difficulties
* Pregnant or breastfeeding
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of significant hematological abnormality or current acute or chronic clinically significant abnormality
* Abnormal serum chemistry laboratory value at Screening deemed to be clinically significant by the Investigator
* Clinically significant cardiovascular disease or abnormal electrocardiogram assessments
* Pre-existing or current signs or symptoms of respiratory failure
* Concurrent acute or chronic clinically significant immunologic, hepatobiliary, or endocrine disease and/or other unstable or major disease other than probable AD or MCI-AD
* Diagnosis of cancer (excluding basal cell carcinoma, squamous cell carcinoma, or prostate carcinoma in situ [Stage 1]) within the past 2 years or a previous (>2 years) diagnosis of cancer that has required any form of intervention or treatment within the past 2 years
* Prior intolerance or hypersensitivity to methylthioninium (MT)-containing drug or methemoglobinemia induced by MT-containing drug, similar organic dyes, or any of the excipients
* Treatment currently or within 90 days before Baseline with Souvenaid®, clozapine, carbamazepine, primidone, valproate, or drugs for which there is a warning or precaution in the labeling about methemoglobinemia at approved doses
* Current or prior participation in any clinical trial of TRx0237; a clinical trial of a product for cognition prior to Baseline in which the last dose was received within 90 days prior to Baseline unless confirmed to have been randomized to placebo; or a clinical trial of any other investigational drug, biologic, device, or medical food in which the last dose was received within 28 days prior to Baseline

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (60):
  - Xenoscience, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Imaging Endpoints Research, Scottsdale, Arizona
  - Atria Clinical Research, Little Rock, Arkansas
  - ATP Clinical Research, Inc., Costa Mesa, California
  - HB Clinical Trials Inc., Fountain Valley, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Excell Research, Inc., Oceanside, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Medical Group, Sherman Oaks, California
  - Visionary Investigators Network, Aventura, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - MD Clinical, Hallandale, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Merrit Island Medical Research, Merritt Island, Florida
  - Health Care Family Rehab and Research, Miami, Florida
  - Optimus Clinical Research, Miami, Florida
  - Biomed Research Institute, Inc, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Bioclinica Research, Orlando, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - The Roskamp Institute, Inc., Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - Advanced Memory Research of NJ PC, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - UBMD Neurology, Buffalo, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Neuroscience Research Center, LLC, Canton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Neurology Diagnostics Inc., Dayton, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - Neural Net Research, Portland, Oregon
  - CBRI - Roper Hospital, Charleston, South Carolina
  - Coastal Neurology, Port Royal, South Carolina
  - Re:Cognition Health, Fairfax, Virginia
  - Kingfisher Cooperative, LLC, Spokane, Washington
  - Universal Research Group, LLC, Tacoma, Washington
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Canada (4):
  - Okanagan Clinical Trials, Ltd., Kelowna, British Columbia
  - Memory Clinic (Ottawa), Ottawa, Ontario
  - Clinique Mémoire de l'Outaouais, Gatineau, Quebec
  - Alpha Recherche Clinique, Québec
- France (9):
  - CHU Bordeaux - Pellegrin, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU de Limoges, Limoges
  - Timone Adults Hospital, Marseille
  - Guidechauliac Hospital, Montpellier
  - Hôpital Laënnec - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CRC Gerontopole Cite de la Sante, Hôpital La Grave, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Italy (9):
  - IRCCS Centro S. Giovanni di Dio Fatebenefratelli, Brescia
  - Foundation Institute G.Giglio, Cefalù
  - Azienda Ospedaliera San Gerardo - Clinica Neurologica, Monza
  - Istituto Neurologico Casimiro Mondino, IRCCS, Pavia
  - University of Perugia, Ospedale S.M. della Misericordia, Perugia
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma
  - IRCCS Fondazione Santa Lucia, Rome
  - Clinica Neurologica Santa Maria della Misericordia, Udine
- Poland (7):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Indywidualna Praktyka Lekarska, Lublin
  - NZOZ Neuro-Kard, Poznan
  - Euromedis Sp. z o.o., Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
- Spain (8):
  - Hospital General de Catalunya, Barcelona
  - Hospitales de Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario QuironSalud Madrid, Madrid
  - Centro de salud de San Juan, Unidad de Investigación Neurociencias, Salamanca
  - Hospital Virgen de la Macarena, Seville
  - Hospital Universitario Mutua Terrassa, Terrassa
  - Hospital Universitario Doctor Peset, Valencia
- United Kingdom (5):
  - Re:Cognition Health, Birmingham
  - Glasgow Memory Clinic Ltd, Glasgow
  - Re:Cognition Health, Guildford
  - Re:Cognition Health - Central London, London
  - Re:Cognition Health, Plymouth

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control: Oral placebo tablets (some of which contain a urinary discolorant) administered twice daily during the double-blind phase, then switched to TRx0237 16 mg/day during the open-label phase
- TRx0237 8 mg/Day: TRx0237 8 mg/day: Oral TRx0237 4-mg tablet administered twice daily during the double-blind phase, then switched to TRx0237 16 mg/day during the open-label phase
- TRx0237 16 mg/Day: TRx0237 16 mg/day: Oral TRx0237 4-mg tablets administered twice daily during the double-blind phase, continued on TRx0237 16 mg/day during the open-label phase
Period: Double-blind Phase
Arm/Group | Control | TRx0237 8 mg/Day | TRx0237 16 mg/Day
Started | 266 | 80 | 252
Completed | 215 | 61 | 194
Not Completed | 51 | 19 | 58
Period: Open-label Phase (All TRx0237 16 mg/Day)
Arm/Group | Control | TRx0237 8 mg/Day | TRx0237 16 mg/Day
Started (14 subjects completed an earlier version of the study protocol, in which there was no open-label phase following the double-blind phase.) | 205 | 57 | 194
Completed | 176 | 47 | 168
Not Completed | 29 | 10 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | TRx0237 8 mg/Day | TRx0237 16 mg/Day | Total
Number analyzed (Participants) | 266 | 80 | 252 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.3) | 71.8 (8.1) | 71.9 (8.6) | 72.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 49 | 161 | 363
  Male | 113 | 31 | 91 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 10 | 2 | 8 | 20
  White | 239 | 73 | 215 | 527
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 16 | 3 | 27 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog11) (16 mg/Day vs Control)
Description: This primary outcome measure was assessed in the TRx0237 16 mg/day group compared to the control group. The scores on this scale range from 0 to 70, with higher numbers indicating a worse outcome (greater impairment).
Time Frame: 52 weeks
Population: Data analyzed using the E-MITTv5 Population, which includes all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline efficacy assessment; results reported for subjects in this population with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline ADAS-cog11 as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 198 | 189
score on a scale | 1.71 [0.69 to 2.73] | 1.34 [0.32 to 2.36]

2. Primary Outcome: Change From Baseline on Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) (16 mg/Day vs Control)
Description: This primary outcome measure was assessed in the TRx0237 16 mg/day group compared to the control group. The scores on this scale range from 0 to 78, with higher numbers indicating a better outcome (lower impairment).
Time Frame: 52 weeks
Population: Data analyzed using the E-MITTv5 Population, which includes all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline efficacy assessment; results reported for subjects in this population with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline ADCS-ADL23 as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 204 | 191
score on a scale | -0.77 [-2.32 to 0.78] | -0.62 [-2.19 to 0.95]

3. Primary Outcome: Number of Study Participants With Serious and Non-serious Adverse Events (16 mg/Day vs Control)
Description: This primary outcome measure was assessed in the TRx0237 16 mg/day group compared to the placebo group. All laboratory test or vital sign parameter abnormalities deemed clinically significant by the Investigator are to be reported as adverse events.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 266 | 252
Participants
  Number of study participants with serious adverse events | 17 | 18
  Number of study participants with non-serious adverse events | 146 | 131

4. Secondary Outcome: Change in Annualized Rate of Whole Brain Atrophy (16 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 16 mg/day group compared to the control group.
Time Frame: 52 weeks
Population: Data analyzed using the MI-MITTv5 Population, which includes all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline MRI assessment; results reported for subjects in this population with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline MRI whole brain volume as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: mm3/year
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 175 | 165
mm3/year | -11137.44 [-12682.86 to -9592.01] | -11162.70 [-12711.43 to -9613.98]

5. Secondary Outcome: Change in Standardized Uptake Value Ratio (SUVR) Based on Temporal Lobe 18F-fluorodeoxyglucose Positron Emission Tomography (18F-FDG-PET) (16 mg/Day vs Control)
Description: This secondary outcome measure (normalized to pons) was assessed in the TRx0237 16 mg/day dose group compared to the control group, and restricted to subjects with Clinical Dementia Rating (CDR) 0.5 at Screening.
Time Frame: 52 weeks
Population: Data analyzed using the PI-MITTv5 Population, which includes all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline 18F-FDG-PET SUVR assessment; results reported for subjects with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (ANCOVA with fixed effects, including Baseline PET temporal lobe glucose uptake as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 88 | 93
ratio | -0.025 [-0.036 to -0.015] | -0.026 [-0.036 to -0.016]

6. Secondary Outcome: Change in Annualized Rate of Temporoparietal Lobe Atrophy (16 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 16mg/day group compared to the control group.
Time Frame: 52 weeks
Population: Data analyzed using the MI-MITTv5 Population (all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline MRI assessment); results reported for subjects in this population with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline MRI whole temporoparietal lobe volume as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: mm3/year
Arm/Group | Control | TRx0237 16 mg/Day
Number analyzed (Participants) | 175 | 165
mm3/year | -740.79 [-821.39 to -660.19] | -711.14 [-791.96 to -630.32]

7. Secondary Outcome: Change From Baseline on Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog11) (8 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 8 mg/day group compared to the control group. The scores on this scale range from 0 to 70, with higher numbers indicating a worse outcome (greater impairment).
  Note: Estimates for the Control Arm in the primary outcome and this secondary outcome are estimated using separate Mixed Models for Repeated Measures (MMRM). Thus, it is appropriate for the two models to yield two slightly different estimates for the Control Arm change as the comparator is different in each case and the model uses this information to make its estimates.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- TRx0237 8 mg/Day: TRx0237 8 mg/day: Oral TRx0237 4-mg tablets administered twice daily
Arm/Group | Control | TRx0237 8 mg/Day
Number analyzed (Participants) | 198 | 47
score on a scale | 1.78 [0.79 to 2.77] | 1.06 [-0.89 to 3.01]

8. Secondary Outcome: Change From Baseline on Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) (8 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 8 mg/day group compared to the control group. The scores on this scale range from 0 to 78, with higher numbers indicating a better outcome (lower impairment).
  Note: Estimates for the Control Arm in the primary outcome and this secondary outcome are estimated using separate Mixed Models for Repeated Measures (MMRM). Thus, it is appropriate for the two models to yield two slightly different estimates for the Control Arm change as the comparator is different in each case and the model uses this information to make its estimates.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | TRx0237 8 mg/Day
Number analyzed (Participants) | 204 | 47
score on a scale | -0.82 [-2.36 to 0.72] | -1.41 [-4.46 to 1.64]

9. Secondary Outcome: Change in Standardized Uptake Value Ratio (SUVR) Based on Temporal Lobe 18F-fluorodeoxyglucose Positron Emission Tomography (18F-FDG-PET) (8 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 8mg/day dose group compared to the control group, and restricted to subjects with Clinical Dementia Rating (CDR) 0.5 at Screening.
  Note: Estimates for the Control Arm in the TRx0237 16 mg/day dose group comparison and this secondary outcome are estimated using separate Mixed Models for Repeated Measures (MMRM). Thus, it is appropriate for the two models to yield two slightly different estimates for the Control Arm change as the comparator is different in each case and the model uses this information to make its estimates.
Time Frame: 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Control | TRx0237 8 mg/Day
Number analyzed (Participants) | 88 | 22
ratio | -0.027 [-0.038 to -0.016] | -0.022 [-0.041 to -0.002]

10. Secondary Outcome: Change in Annualized Rate of Temporoparietal Lobe Atrophy (8 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 8 mg/day dose group compared to the control group.
  Note: Estimates for the Control Arm in the TRx0237 16 mg/day dose group comparison and this secondary outcome are estimated using separate Mixed Models for Repeated Measures (MMRM). Thus, it is appropriate for the two models to yield two slightly different estimates for the Control Arm change as the comparator is different in each case and the model uses this information to make its estimates.
Time Frame: 52 weeks
Population: Data analyzed using the MI-MITTv5 Population (all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug and have a Baseline and at least one valid postbaseline MRI assessment); results reported for subjects in this population with Baseline and Week 52 data. Change from Baseline to Week 52 is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline MRI whole temporoparietal volume as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: mm3/year
Arm/Group | Control | TRx0237 8 mg/Day
Number analyzed (Participants) | 175 | 45
mm3/year | -729.55 [-806.00 to -652.09] | -651.28 [-799.33 to -503.24]

11. Secondary Outcome: Change From Open-Label Baseline on Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog11)
Description: This secondary outcome measure was assessed for the open-label period of the study comparing subjects originally randomized to placebo to subjects originally randomized to either dose of TRx0237. The scores on this scale range from 0 to 70, with higher numbers indicating a worse outcome (greater impairment).
  Note: It was prespecified to combine subjects who received TRx0237 8 mg/day or TRx0237 16 mg/day in the double-blind phase as early starters; thus these are combined for this comparison.
Time Frame: 104 weeks
Population: Data analyzed using the ITTv5-OL Population, which includes all subjects randomized to Protocol Version 5.0+ who received at least one dose of study drug in the open-label (OL) phase; results reported for subjects in this population with a Baseline-OL value and Week 104 data (52 weeks of OL drug). Change from Baseline-OL to Week 104 (52 weeks) is included in the LSM calculation (restricted maximum likelihood-based MMRM with fixed effects, including Baseline-OL ADAS-cog11 as a covariate).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Control to TRx0237 16 mg/Day: Subjects who were randomized to the control arm in the double-blind phase and switched to TRx0237 16 mg/day in the open-label phase (late starters)
- TRx0237 (Either Dose) to TRx0237 16 mg/Day: Subjects who were randomized to the TRx0237 8 mg/day or TRx0237 16 mg/day arms in the double-blind phase and then TRx0237 16 mg/day in the open-label phase (early starters)
Arm/Group | Control to TRx0237 16 mg/Day | TRx0237 (Either Dose) to TRx0237 16 mg/Day
Number analyzed (Participants) | 146 | 179
score on a scale | 2.98 [2.01 to 3.95] | 3.58 [2.70 to 4.47]

12. Secondary Outcome: Number of Study Participants With Serious and Non-serious Adverse Events (8 mg/Day vs Control)
Description: This secondary outcome measure was assessed in the TRx0237 8 mg/day group compared to the control group over 52 weeks. All laboratory test or vital sign parameter abnormalities deemed clinically significant by the Investigator were to be reported as adverse events.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | TRx0237 8 mg/Day
Number analyzed (Participants) | 266 | 80
Participants
  Number of study participants with serious adverse events | 17 | 6
  Number of study participants with nonserious adverse events | 146 | 47

13. Secondary Outcome: Number of Study Participants With Serious and Non-serious Adverse Events (Open-label)
Description: This secondary outcome measure was assessed for all subjects receiving TRx0237 in the open-label phase of the study (in which subjects had received TRx0237 for up to 104 weeks).
  Note: Subjects who received TRx0237 8 mg/day or TRx0237 16 mg/day arms in the double-blind phase are combined for this comparison as all had previously received TRx0237 as compared to those subjects in the control arm who were receiving TRx0237 for the first time in the open-label phase.
Time Frame: 104 weeks
Population: A total of 7 subjects had discontinued study drug in the double-blind phase but completed this phase and continued to attend study visits in the open-label (OL) phase off-treatment. As these subjects did not receive TRX0237 16 mg/day in the OL phase, they are not included in the OL-Safety Population (N=449) and thus are not included in these comparisons.
Measure: Count of Participants; unit: Participants
Groups:
- Control to TRx0237 16 mg/Day: Subjects who were randomized to the control arm in the double-blind phase and switched to TRx0237 16 mg/day in the open-label phase
- TRx0237 (Either Dose) to TRx0237 16 mg/Day: Subjects who were randomized to the TRx0237 8 mg/day or TRx0237 16 mg/day arms in the double-blind phase and then received TRx0237 16 mg/day in the open-label phase
Arm/Group | Control to TRx0237 16 mg/Day | TRx0237 (Either Dose) to TRx0237 16 mg/Day
Number analyzed (Participants) | 201 | 248
Participants
  Number of study participants with serious adverse events | 14 | 13
  Number of study participants with nonserious adverse events | 88 | 101

ADVERSE EVENTS:
Time Frame: 104 weeks (2 years)
Description: AEs were ascertained at each study visit by asking the subject and study partner how the subject had been since the last visit. Additionally, AEs were also reported based on study safety assessments performed at each study visit.
Groups:
- Double-blind Control: Control: Oral placebo tablets (some of which contain a urinary discolorant) administered twice daily
- Double-blind TRx0237 8 mg/Day: TRx0237 8 mg/day: Oral TRx0237 4-mg tablet administered twice daily
- Double-blind TRx0237 16 mg/Day: TRx0237 16 mg/day: Oral TRx0237 4-mg tablets administered twice daily in the double-blind phase
- Open-label TRx0237 16 mg/Day: TRx0237 16 mg/day: Oral TRx0237 4-mg tablets administered twice daily in the open-label phase (all subjects who completed the double-blind phase and entered the open-label phase transitioned to receive this treatment)
Arm/Group | Double-blind Control | Double-blind TRx0237 8 mg/Day | Double-blind TRx0237 16 mg/Day | Open-label TRx0237 16 mg/Day
All-Cause Mortality (participants affected / at risk) | 1/266 | 0/80 | 1/252 | 8/449
Serious Adverse Events (participants affected / at risk) | 17/266 | 6/80 | 18/252 | 27/449
Other Adverse Events (participants affected / at risk) | 30/266 | 12/80 | 22/252 | 40/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Control (N=266) | Double-blind TRx0237 8 mg/Day (N=80) | Double-blind TRx0237 16 mg/Day (N=252) | Open-label TRx0237 16 mg/Day (N=449)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Lens discolouration (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gait inability (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Neuropsychiatric symptoms (Psychiatric disorders) | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Control (N=266) | Double-blind TRx0237 8 mg/Day (N=80) | Double-blind TRx0237 16 mg/Day (N=252) | Open-label TRx0237 16 mg/Day (N=449)
Corona virus infection (Infections and infestations) | 11 | 6 | 7 | 18
Fall (Injury, poisoning and procedural complications) | 11 | 2 | 5 | 15
Headache (Nervous system disorders) | 8 | 5 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT03446001/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03446001/SAP_002.pdf